CLINICAL TRIAL: NCT07158593
Title: Universal Prevention Program "Claudia Carraro" for Improving Body Image and Promoting Healthy Lifestyles in Adolescent Boys and Girls: a Cluster Randomized Controlled Trial With 24-week Follow-up
Brief Title: School-Based Eating Disorder Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Villa Garda Hospital (Other)
Responsible Party: Principal Investigator, Riccardo Dalle Grave, Head of Nutrition and Endocrinology at Villa Garda Hospital, Villa Garda Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2505CESC
Record Dates: First submitted 2025-08-28; First posted 2025-09-08 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Prevention Program; Wait List Control
Keywords: eating disorders; adolescents; cognitive behavior therapy; universal prevention program; risk factors; school-based interventions
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention arm, includes studed who attended the "Claudia Carraro" prevention program. It is grounded in a cognitive-behavioral conceptualization of the development of eating disorders or disordered eating. The program was designed to address specific and non-specific risk factors that appear relevant: body dissatisfaction and unhealthy weight control behaviors. Its dual objective is to help participants reduce the importance they place on body weight and shape in self-evaluation while simultaneously promoting healthy weight regulation through adherence to Mediterranean dietary guidelines and an active lifestyle.
  The strategies and procedures used are derived from cognitive behavioral therapy protocols for eating disorders (Dalle Grave & Calugi, 2020). The intervention is delivered by psychologists specialized in eating and weight disorders using an interactive, rather than didactic, format, involving small group activities and assigned homework tasks between sessions.
  Interventions: Other: Claudia carraro prevention program
- Control (No Intervention): No intervention. The control group received the intervention after the 24 weeks

INTERVENTIONS:
Other: Claudia carraro prevention program — The "Claudia Carraro" prevention program is grounded in a cognitive-behavioral conceptualization of the development of eating disorders or disordered eating. The program was designed to address specific and non-specific risk factors that appear relevant: body dissatisfaction and unhealthy weight control behaviors. Its dual objective is to help participants reduce the importance they place on body weight and shape in self-evaluation while simultaneously promoting healthy weight regulation through adherence to Mediterranean dietary guidelines and an active lifestyle.
  The strategies and procedures used are derived from cognitive behavioral therapy protocols for eating disorders (Dalle Grave & Calugi, 2020). The intervention is delivered by psychologists specialized in eating and weight disorders using an interactive, rather than didactic, format, involving small group activities and assigned homework tasks between sessions.
  Arms: Intervention

SUMMARY:
This is a cluster randomized controlled trial with two assessment points (baseline and 24-week follow-up) comparing the Claudia Carraro prevention program to a no-intervention control group. The intervention group was also assessed at post-intervention. To ensure that all students benefit from the intervention, the control group received the intervention after the 24 weeks.

Randomization was performed at the school level, not the student level.

DETAILED DESCRIPTION:
Participants were recruited from January 2020 and December 2024. Secondary school administrators were contacted via telephone and/or email and provided with a letter outlining the core principles of the prevention program. If the school principal (or a designated representative) agreed to participate, they were asked to sign a formal agreement to take part in the intervention.

Students in the first or second year of upper secondary school and those who signed a written informed consent were included. Also, the informed consent should be signed by their parents. However, were excluded from the study students who self-reported diagnosis of an ED (these individuals could participate in the intervention but were excluded from data analysis).

Theoretical Framework The "Claudia Carraro" prevention program is grounded in a cognitive-behavioral conceptualization of the development of eating disorders or disordered eating. The program was designed to address specific and non-specific risk factors that appear relevant: body dissatisfaction and unhealthy weight control behaviors. Its dual objective is to help participants reduce the importance they place on body weight and shape in self-evaluation while simultaneously promoting healthy weight regulation through adherence to Mediterranean dietary guidelines and an active lifestyle.

The strategies and procedures used are derived from cognitive behavioral therapy protocols for eating disorders (Dalle Grave & Calugi, 2020). The intervention is delivered by psychologists specialized in eating and weight disorders using an interactive, rather than didactic, format, involving small group activities and assigned homework tasks between sessions.

Facilitator Training and Supervision Facilitators received formal training through a one-day seminar conducted by the principal and co-investigators. To assess adherence to the intervention protocol, all sessions were audio-recorded, and the program coordinators reviewed a random sample.

Facilitators were selected based on documented expertise in eating disorders and cognitive-behavioral therapy.

Program Structure The program consists of three sessions, each lasting 2.5 hours, delivered over three consecutive weeks. Each session builds on the previous one and begins with a review of key concepts and skills. Sessions involve interactive teaching, slide presentations, group work, and homework assignments to be completed between meetings. See Table 1 for an overview of the activities.

Measures Case Report Form (CRF) The CRF, to be completed by each participant, included general demographic and anthropometric data (date of birth, weight, height, gender) and two screening questions regarding the presence or being in treatment for an eating disorder.

Self-report Questionnaires Eating Disorder Examination Questionnaire (EDE-Q) (Calugi et al., 2017; Fairburn et al., 2008): A validated Italian version that assesses the severity of eating disorder psychopathology over the past 28 days. The EDE-Q assesses eating disorder psychopathology with a global score and four subscales (restraint, eating concern, weight concern, shape concern) and eating disorder behaviours (objective binge-eating, self-induced vomiting, laxative misuse, excessive exercise).

Short Form of the International Physical Activity Questionnaire (IPAQ-SF) (Craig et al., 2003; Mannocci et al., 2010): A validated Italian questionnaire assessing self-reported physical activity across four domains: walking, moderate-intensity activity, vigorous-intensity activity, and time spent sitting.

Mediterranean Diet Adherence Questionnaire (QueMD) (Gnagnarella et al., 2018): A validated Italian-language instrument measuring adherence to the Mediterranean diet.

Questionnaire Administration Timeline Baseline: Administered approximately 30 minutes before the first intervention session (if permitted by the school) or during the first 30 minutes of the session itself in participants allocated to the intervention. Administered about 24 weeks before the intervention in participants allocated to the control group. All questionnaires were collected immediately after completion.

Post-intervention: Administered and collected during the final 30 minutes of the third (final) intervention session (only in participants who attended the intervention).

24-week follow-up: Administered during a dedicated 30-minute session held 24 weeks after the intervention in participants allocated to the intervention. Administered after 24 weeks from the baseline and corresponding to the first intervention session in participants allocated to the control group.

All informed consent forms and data privacy agreements were collected by the professional responsible for delivering the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Students in the first or second year of upper secondary school
* Students who signed a written informed consent
* Informed consent signed by their parents

Exclusion Criteria:

* Students who self-reported diagnosis of an eating disorder (these individuals could participate in the intervention but were excluded from data analysis)

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1205 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Examination Questionnaire | Baseline and 24-week follow-up. The intervention group was also assessed at post-intervention
  The Eating Disorder Examination Questionnaire (EDE-Q) (Calugi et al., 2017; Fairburn et al., 2008) is a validated Italian version that assesses the severity of eating disorder psychopathology over the past 28 days. The EDE-Q assesses eating disorder psychopathology with a global score and four subscales (restraint, eating concern, weight concern, shape concern) and eating disorder behaviours (objective binge-eating, self-induced vomiting, laxative misuse, excessive exercise). Scores range from 0 to 6. Higher scores indicate higher eating disorder psychopathology.

SECONDARY OUTCOMES:
Short Form of the International Physical Activity Questionnaire | Baseline and 24-week follow-up. The intervention group was also assessed at post-intervention
  The Short Form of the International Physical Activity Questionnaire (IPAQ-SF) (Craig et al., 2003; Mannocci et al., 2010) is a validated Italian questionnaire assessing self-reported physical activity across four domains: walking, moderate-intensity activity, vigorous-intensity activity, and time spent sitting. Scores are categorized as follow: Low Activity (<600 MET-min/week), Moderate Activity (600-2999 MET-min/week), and High Activity (≥3000 MET-min/week).
Mediterranean Diet Adherence Questionnaire | Baseline and 24-week follow-up. The intervention group was also assessed at post-intervention
  The Mediterranean Diet Adherence Questionnaire (QueMD) (Gnagnarella et al., 2018) is a validated Italian-language instrument measuring adherence to the Mediterranean diet. The score ranges from a minimum of 0 to a maximum of 9, with higher scores indicating greater adherence to the Mediterranean diet.

CONTACTS AND LOCATIONS:
Locations (1):
- Villa Garda Hospital, Verona, Veneto, Italy